CLINICAL TRIAL: NCT05780970
Title: Exploring the Familial Reach of Adolescent Obesity Treatment
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Connecticut (Other); University of North Carolina (Other); University of Tennessee (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM20014304 Phase 3; R21HD105906 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Obesity
Keywords: Pediatric Obesity; Lifestyle Intervention; Family-Level Change; Family-based Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-targeted individuals: Non-targeted children and caregivers living in the same household as the target parent/adolescent dyad. Non-targeted meaning they did not receive the TEENS+ intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Non-treated children and caregivers complete assessments only. The primary (treated) parent / adolescent dyad participate in family based weight management treatment through the main trial. In the main trial, families are randomized to either TEENS+Parents as Coaches (parent skills training) or TEENS+Parent Weight Loss (parent behavioral weight loss).

SUMMARY:
An observational study ancillary to the randomized clinical trial (RCT) TEENS+ (R01HD095910), a family-based lifestyle intervention, for adolescents with obesity, to determine: 1) if family-wide changes to the shared home environment are implemented, 2) if ripple effects to untreated family members are observed, and 3) whether these changes are predictive of adolescents' weight management success.

Funding support from NIH via R21HD105906.

DETAILED DESCRIPTION:
Investigators will recruit non-targeted children (8-17yrs) and caregivers living in the same household as the target TEENS+ parent/adolescent dyad. At 0, 2, 4 and 8m, the target adolescent/parent dyad (n=60), and non-targeted children and caregivers will complete anthropometric assessments, and measures of the shared home feeding and weight-related environment will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Untreated children: must be between 8-17 years of age and primarily living in the same household as the TEENS+ participants.
* Untreated caregiver: must be 18 years of age or older and primarily living in the same household as the TEENS+ participants.
* Treated caregivers: must have another individual in the household that meets the eligbility for an untreated child or untreated caregiver.

Exclusion Criteria:

* temporarily (<1yr) living in the home
* children with a BMI<5th%ile or caregivers with a BMI<18.5 kg/m2
* non-English speaking
* medical condition(s) that may be associated with unintentional weight change or significant disruption to eating behaviors (e.g., hypothalamic injury, Prader-Willi, G-tube placement, or malignancy
* clinically significant eating disorder (e.g., anorexia nervosa or bulimia nervosa)
* following a medically-supervised/prescribed diet
* psychiatric, cognitive, physical or developmental conditions that would impair the individual's ability to complete assessments.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals residing in the home with the parent/child dyad who are participating in the TEENS+ (R01HD095910) RCT. Participating dyads must have overweight or obesity.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Family-level changes to the shared home environment. | 4 months (baseline to 4 months)
  Changes in the home food available and the home exercise and electronic media environment.
Weight changes. | 4 months (baseline to 4 months)
  Weight changes observed among untreated individuals (child zBMI and caregiver % weight loss)
Household changes and target adolescent weight. | 8 months [weight loss (baseline to 4 months) and maintenance (4-8)]
  Associations between household changes and target adolescent weight loss and maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Bean, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States

REFERENCES:
- [Derived] Brown KL, LaRose JG, Raynor HA, Gorin AA, Thornton LM, Farthing S, Tatum K, Bean MK. Study design and rationale for TEENS+REACH: Evaluating ripple effects of a family-based lifestyle intervention to untreated family members. Contemp Clin Trials Commun. 2024 Feb 15;38:101276. doi: 10.1016/j.conctc.2024.101276. eCollection 2024 Apr. PMID 38404649

DOCUMENTS (1):
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT05780970/ICF_000.pdf